CLINICAL TRIAL: NCT03214484
Title: A Prospective Study Comparing the Evolution of Visual Acuity Measured by Electronic Tablet or Computer and the Visual Acuity Measured by ETDRS in Patients Monitored and Treated for Exudative AMD
Brief Title: The Evolution of Visual Acuity Measured by Electronic Tablet / Computer of Exudative AMD Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Principal Investigator, Frédéric QUEGUINER, MD, Ophtalmologist Principal Investigator, Hospital St. Joseph, Marseille, France
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Sight Study
Record Dates: First submitted 2017-05-31; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Macular Degeneration Exudative Eye Bilateral

STUDY DESIGN:
Intervention Model Description: In total, 80 patients (40 for the Electronc Tablet group, 40 for the computeur group) will be included in the study.
  Using the pre-established randomization list, in order of inclusion in the study, each patient will be assigned to one of the 2
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- electronc tablet (Active Comparator): On ET or Computer, the AV is measured at a closer distance (40 cm and 80 cm, respectively). At this closer distance (ie near and near vision), the eccentric fixation is much more Difficult to perform, unnatural, often requiring learning in the context of low vision rehabilitation.
  Our aim is to compare the evolution curves of the Visual Acuity (AV) measured in each patient on Electronic Tablet (TE)/ computer(O) and on the Early Treatment of Diabetic Retinopathy Study (ETDRS) scale, in order to check the reliability of the measurements performed by TE / O by comparing them with a well-known reference measure And is routinely practiced routinely in ophthalmology centers.
  Interventions: Other: By comparing the evolution of the visual acuity curves.; Other: By comparing the evolution of the curves.
- computer (Active Comparator): On ET or Computer, the AV is measured at a closer distance (40 cm and 80 cm, respectively). At this closer distance (ie near and near vision), the eccentric fixation is much more Difficult to perform, unnatural, often requiring learning in the context of low vision rehabilitation.
  Our aim is to compare the evolution curves of the Visual Acuity (AV) measured in each patient on Electronic Tablet (TE)/ computer(O) and on the Early Treatment of Diabetic Retinopathy Study (ETDRS) scale, in order to check the reliability of the measurements performed by TE / O by comparing them with a well-known reference measure And is routinely practiced routinely in ophthalmology centers.
  Interventions: Other: By comparing the evolution of the visual acuity curves.; Other: By comparing the evolution of the curves.

INTERVENTIONS:
Other: By comparing the evolution of the visual acuity curves. — By comparing the evolution of the curves, the investigator can confirm that the AV measured on ET / Computer can be an interesting and useful element to help us follow up our patients and improve the quality of life's patients by decreasing the number of visits control.
Other: By comparing the evolution of the curves. — By comparing the evolution of the curves, the investigator can confirm that the AV measured on ET / Computer can be an interesting and useful element to help us follow up our patients and improve the quality of life's patients by decreasing the number of visits control.

SUMMARY:
This pathology, DMLA, whose evolution is chronic, requires regular follow-up and care (IVTs) over a long period (several months or even years).

Increasing the number of patients to be followed and treated poses increasing problems for ophthalmologists to ensure regular follow-up of patients, followed by a need for satisfactory functional results.

Moreover, this regular follow-up imposes enormous constraints on patients and their families (some children or patients are still working).

Studies are beginning to emerge on the reliability of patient follow-up in telemedicine. The use of a measure of visual acuity by patients, Electronic Tablet (TE) or computer (O), and at home, seems a logical step to help us improve the quality of patient follow-up while spacing controls.

The aim of our study is thus to demonstrate that the measurement of the VA performed by TE or O is reliable. Indeed, during the follow-up of the patients, in the case where the patient's AV decreases, and whatever the reason

DETAILED DESCRIPTION:
Our aim is to compare the evolution curves of the Visual Acuity (AV) measured in each patient on Electronic Tablet (TE)/ computer(O) and on the Early Treatment of Diabetic Retinopathy Study (ETDRS) scale, in order to check the reliability of the measurements performed by TE / O by comparing them with a well-known reference measure And is routinely practiced routinely in ophthalmology centers.

Measurement of visual acuity on TE / O will be carried out on an ETDRS AV scale, the size of the letters having been adapted to the reading distance (80 cm by 0.40 cm on the tablet). An ETDRS intermediate vision (EVI) or meadow vision (TEU) score according to the group will be established in the same way. The VA measurement will be supervised by a CRA trained to the extent of the VA, without the orthoptist or ophthalmologist being informed of the results obtained.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over 50 years of age.
* Patient monitored and treated in the department by intravitreal injections of anti VEGF (aflibercept or ranibizumab) in the indication of treatment.
* Patient with exudative AMD
* Patient who consented to participate in the study
* Patient who is able to understand the study and use a TE / O
* Patient with AV greater than or equal to 20/100
* Patient affiliated to a health

Exclusion Criteria:

* Patient having expressed his / her refusal on the collection of the medical data of his file at the end of the study
* Patient treated with non-AMD pathology
* Patient with AV less than 20/100
* Vulnerable person: protected by the law: guardianship, curatorship.
* Person participating in another test

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-06-02 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | Day 0
  Visual acuity will be evaluated by Electronic Tablet (TE) and Early Treatment of Diabetic Retinopathy Study (ETDRS scale) for the first group of patients, and by computer (O) and ETDRS for the second group of patients.
Visual acuity | Month 1
  Visual acuity will be evaluated by Electronic Tablet (TE) and Early Treatment of Diabetic Retinopathy Study (ETDRS scale) for the first group of patients, and by computer (O) and ETDRS for the second group of patients.
Visual acuity | Month 2
  Visual acuity will be evaluated by Electronic Tablet (TE) and Early Treatment of Diabetic Retinopathy Study (ETDRS scale) for the first group of patients, and by computer (O) and ETDRS for the second group of patients.
Visual acuity | Month 3
  Visual acuity will be evaluated by Electronic Tablet (TE) and Early Treatment of Diabetic Retinopathy Study (ETDRS scale) for the first group of patients, and by computer (O) and ETDRS for the second group of patients.
Visual acuity | Month 4
  Visual acuity will be evaluated by Electronic Tablet (TE) and Early Treatment of Diabetic Retinopathy Study (ETDRS scale) for the first group of patients, and by computer (O) and ETDRS for the second group of patients.
Visual acuity | Month 5
  Visual acuity will be evaluated by Electronic Tablet (TE) and Early Treatment of Diabetic Retinopathy Study (ETDRS scale) for the first group of patients, and by computer (O) and ETDRS for the second group of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Saint Joseph, Marseille, France

IPD SHARING:
Plan to Share IPD: No